CLINICAL TRIAL: NCT02150681
Title: MBCT for Perinatal Women With Mood Disorders
Brief Title: Mindfulness-Based Cognitive Therapy for Perinatal Women With Mood Disorders
Acronym: MBCT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: University of Colorado, Boulder (Other)
Responsible Party: Principal Investigator, David J. Miklowitz, Ph.D., Professor of Psychiatry, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-003212
Record Dates: First submitted 2014-05-27; First posted 2014-05-30 (Estimated); Last update posted 2014-05-30 (Estimated); Status verified 2014-05

CONDITIONS: Major Depressive Disorder; Bipolar Disorder
Keywords: preconception; pregnancy; postpartum; women
MeSH Terms: conditions — Depressive Disorder, Major; Bipolar Disorder | interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mindfulness-based cognitive therapy (Experimental): 8 class sessions of mindfulness therapy given in a group setting, with one 2-hr session per week for 8 weeks.
  Interventions: Behavioral: Mindfulness-based cognitive therapy

INTERVENTIONS:
Behavioral: Mindfulness-based cognitive therapy — This is an 8-week treatment for women with mood disorders. The focus of sessions 1 through 4 is to establish a foundation of mindfulness practice and bringing nonjudgmental awareness to the present moment, beginning with concrete targets of attention and moves to more emotionally challenging and abstract targets (e.g., depression-specific thoughts). Participants are guided to become aware of the automatic patterns of their minds and in such moments to return attention to thoughts, feelings and body sensations. Participants engage experientially with the ways in which thoughts and emotions become engaged with rumination. In sessions 5 through 8, participants learn to extend their basic mindfulness skills to become aware of relapse risk signs and develop prevention plans.

SUMMARY:
This study will investigate the effectiveness of mindfulness-based cognitive therapy (MBCT) for mood stabilization in perinatal women (preconception, pregnant, and postpartum) with a history of mood disorders. MBCT is a short-term group psychotherapy that has shown effectiveness in preventing depressive relapse. MBCT teaches mindfulness practices and cognitive-behavioral techniques.

DETAILED DESCRIPTION:
Approximately 10-15% of women experience depression following the birth of a child. Depression during pregnancy is also common. Women with a history of depression or bipolar disorder are at increased risk of depressive relapse or exacerbation of mood symptoms during the perinatal period. Perinatal depression is associated with a host of negative consequences that can affect the mothers, infants, and families. Women with perinatal depression may have trouble with parenting, marital quality, and employment. Children of mothers with perinatal depression may suffer intellectually or emotionally. These children are also more likely to develop a mood disorder or other psychiatric disorders throughout their lifetimes compared to children whose mothers have not been depressed. Prevention efforts during the preconception, pregnancy, and postpartum periods are of considerable public health benefit. However, perinatal women are often reluctant to start or continue psychotropic medications due to concerns about their influence on the developing fetus or nursing infant. Therefore, psychosocial treatments that modify key vulnerability factors, without medication side effects, are likely to be of strong interest to women who might otherwise remain untreated.

This study will investigate the effectiveness of mindfulness-based cognitive therapy (MBCT) for mood stabilization in perinatal women (preconception, pregnant, and postpartum) with a history of mood disorders. MBCT is a short-term group psychotherapy that has shown effectiveness in preventing depressive relapse. MBCT teaches mindfulness practices and cognitive-behavioral techniques. Mindfulness is the practice of cultivating a non-judgmental awareness of internal experiences (thoughts, feelings, and body sensations) and external experiences. Cognitive-behavioral techniques focus on identifying maladaptive thoughts and behaviors before they spiral into a depressive episode. MBCT teaches observational skills and helpful techniques for responding to distorted or dysfunctional thoughts and behaviors, thereby preventing an impending depressive relapse.

The investigators plan to (1) recruit 20 perinatal women at each of two sites with a history of major depressive disorder or bipolar disorder (currently in remission or partial remission), (2) ascertain their diagnoses and eligibility, (3) collect baseline data (e.g., demographic information, mood and anxiety symptoms), and (4) conduct open-trial MBCT groups with 10-12 women in each group. The investigators examine the feasibility of identifying, enrolling, and retaining perinatal women at high risk for mood episodes in an 8-week MBCT group psychotherapy. Treatment effectiveness, acceptability, and satisfaction will be assessed at the end of treatment, at 1 month post-treatment, and 6 months post-treatment.

This study will contribute to the field's understanding of non-pharmacological prevention options for perinatal and postnatal women at risk for mood episode relapse. MBCT could fill an urgently needed gap in services for preconception, pregnant, and postpartum women who are at increased risk for relapse, and who wish to learn efficacious prevention skills. Given the long-term adverse consequences of untreated perinatal mood episodes for women and their children; low rates of treatment seeking; and concerns associated with pharmacological treatments, the development of a viable psychosocial intervention may have significant benefits for women, children, and society at large.

ELIGIBILITY:
Inclusion Criteria:

Eligible women for this study

* will be planning pregnancy within the forthcoming year, are pregnant, or within one year postpartum

  * will meet criteria for at least one prior Diagnostic and Statistical Manual of Mental Disorders, 4th Ed., Revised major depressive, hypomanic, or manic episode,
  * has met lifetime Diagnostic and Statistical Manual criteria for bipolar I, II, or not otherwise specified disorder or major depressive disorder;
  * are available for group intervention scheduled meetings,
  * speak and read English,
  * age 18 or older.

Exclusion Criteria:

* schizophrenia, schizoaffective disorder, or current psychosis;

  * organic mental disorder or pervasive developmental delay
  * current eating disorder;
  * current substance abuse or dependence;
  * imminent suicide or homicide risk;
  * history of violent behaviors toward others;
  * current thoughts of harm to an unborn or recently born child; or
  * currently experiencing a mood episode that meets full Diagnostic and Statistical Manual criteria.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2012-10; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Change in Self-Rated Depression from Pretreatment to Post-treatment to 1- and 6- months post-treatment | Pretreatment to Post-treatment (2 months), 1 month post-treatment, and 6 months post-treatment
  The primary outcome is self-rated Beck Depression Inventory, II scores at the pretreatment baseline and again at Post-treatment (8 weeks), and then at 1- month and 6-months post-treatment

SECONDARY OUTCOMES:
Change in Observer-Rated Depression from Pretreatment to Post-treatment to 1- and 6 months post-treatment | Pretrreatment to Post-treatment; one-month post-treatment and 6-months post-treatment
  Depression will be measured using the Hamilton Rating Scale for Depression at pretreatment, post-treatment, 1 month, and 6 months after the end of mindfulness-based cognitive therapy sessions
Changes in Anxiety Symptoms | Pretreatment to 6 months post-treatment
  Changes in State-Trait Anxiety Inventory, State Scale from baseline to post-treatment, 1 month, and 6 months
Changes in mania symptoms | Pretreatment to 6 months post-treatment
  Changes in Young Mania Rating Scale scores measured at 4 times: pretreatment, post-treatment, 1 month and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: David J. Miklowitz, Ph.D., Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - University of California, Los Angeles, Los Angeles, California
  - University of Colorado, Boulder, Colorado

REFERENCES:
- See also: This organization, which funded this research, provides considerable information on bipolar disorder and mindfulness treatments. — http://albertsfoundation.org